CLINICAL TRIAL: NCT02144545
Title: Study of Impact of the Size of Gastric Sleeve o the Weight Loss in Patients Submitted to Bariatric Surgery. Evaluation of Changes in Gastric Motility and Endocrine-metabolic Function.
Brief Title: Impact of Size of Gastric Sleeve on the Weight Loss. Correlation With Gastric Function and Endocrine-metabolic Changes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-RES-2012-178
Record Dates: First submitted 2013-11-19; First posted 2014-05-22 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Obesity, Morbid
Keywords: Surgery; Morbid Obesity; Bariatric surgery; Sleeve gastrectomy; Bougie Size; Distance from pylorus; Hormones; Gastric remanent
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bougie Size 33Fr Distance pylorus 2 cm (Experimental): Sleeve gastrectomy with a 33Fr bougie size and 2 cm distance from the pylorus.
  Interventions: Procedure: Bougie Size 33 Fr; Procedure: Distance pylorus 2 cm
- Bougie Size 33Fr Distance pylorus 5 cm (Experimental): Sleeve gastrectomy with a 33Fr bougie size and 5 cm distance from the pylorus
  Interventions: Procedure: Bougie Size 33 Fr; Procedure: Distance pylorus 5 cm
- Bougie Size 42Fr Distance pylorus 2 cm (Experimental): Sleeve gastrectomy with a 42Fr bougie size and 2 cm distance from the pylorus
  Interventions: Procedure: Bougie Size 42 Fr; Procedure: Distance pylorus 2 cm
- Bougie Size 42Fr Distance pylorus 5 cm (Experimental): Sleeve gastrectomy with a 42Fr bougie size and 2 cm distance from the pylorus
  Interventions: Procedure: Bougie Size 42 Fr; Procedure: Distance pylorus 5 cm

INTERVENTIONS:
Procedure: Bougie Size 33 Fr — Comparison of the bougie size and distance from the pylorus for the sleeve gastrectomy
  Arms: Bougie Size 33Fr Distance pylorus 2 cm; Bougie Size 33Fr Distance pylorus 5 cm
Procedure: Bougie Size 42 Fr — Comparison of the bougie size and distance from the pylorus for the sleeve gastrectomy
  Arms: Bougie Size 42Fr Distance pylorus 2 cm; Bougie Size 42Fr Distance pylorus 5 cm
Procedure: Distance pylorus 2 cm — Comparison of the bougie size and distance from the pylorus for the sleeve gastrectomy
  Arms: Bougie Size 33Fr Distance pylorus 2 cm; Bougie Size 42Fr Distance pylorus 2 cm
Procedure: Distance pylorus 5 cm — Comparison of the bougie size and distance from the pylorus for the sleeve gastrectomy
  Arms: Bougie Size 33Fr Distance pylorus 5 cm; Bougie Size 42Fr Distance pylorus 5 cm

SUMMARY:
Morbid Obesity (MO) is considered the most important epidemic in the developed world in the twenty-first century. After initial assessment of morbidly obese patients and the exclusion of potentially correctable causes, management involves a combination of dietary changes, cognitive therapy, physical activity, psychological support and pharmacological treatment. However, any combination of these factors has proven long-term effectiveness in achieving significant and sustained reduction of excess weight. Currently, surgery is the only treatment capable of achieving this goal, interacting also with significant improvement in quality of life and overall long-term mortality.

In recent years, several authors have reported excellent short-term results with performing sleeve gastrectomy, but whether some aspects regarding the variability of gastric tubulization design could influence the results obtained in relation to weight loss and functional changes and gastric hormones.

The main objective of this study is to assess the size of the gastric tubulization (based probe calibration and the distance from the pylorus to which initiate gastric section) that can provide a better clinical outcome (such as excess weight loss) in patients undergoing surgery for morbid obesity. Secondary objectives were to assess the morphological changes, physiological and hormonal obtained according to the size of the gastric tubulization and its effect on weight loss patients.

DETAILED DESCRIPTION:
HYPOTHESIS Surgical major factors which determine the size of the gastric pouch after performing a a sleeve gastrectomy are the diameter of the remanent stomach (influenced by the diameter of the bougie size) and the residual antrum.

Whereas gastrectomy is a restrictive procedure, we postulate that the variation of these factors can have a significant impact on clinical outcomes in terms of weight loss and improvement in comorbidities in addition to possible changes in the hormone pattern

OBJECTIVE:

* Primary Outcome Measure:

Weight loss one year after surgery

* Secondary Outcome Measures:
* Morphological changes induced by the size of the gastric tubulization
* Gastric antrum volume
* Gastric body volume
* Correlation between gastric volumes and weight loss
* Gastric emptying
* Hormone levels (before and after surgery) and relation with weight loss
* Quality of life

DATA TO ANALIZE

We will analyze the following key variables:

* BMI (body mass index)
* Preoperative gastric volume
* Postoperative gastric volume. An evaluation of the variation of these data in two stages (one month and one year after surgery) in each patient group and the comparison will be made between groups.

Secondary variables to analyze are:

- Gastric emptying, analyzed in relation to baseline (preoperative)

* Lower esophageal sphincter pressure
* The number of episodes of gastroesophageal reflux, the number of reflux episodes longer than 5 minutes, the percentage of time with pH below 4
* Plasma hormones listed below An evaluation of the temporary modification of these variables to the month and year of surgery in relation to preoperative values in each patient group and the comparison will be made between the four groups.
* Gastric volume study Methodology For the evaluation of the patients an abdominal CT scan in multislice device will be performed. Diluted oral contrast was administered 3% (amidotrizoate meglumine, sodium amidotrizoate Gastrografin ®) for a maximum distension of the stomach or gastric remnant in order to assess gastric volume or its remnant. Cuts will be made within 45 minutes of ingestion of oral contrast and perform a CT without intravenous contrast supine, including from the tracheal carina to pubic symphysis. Cuts are initiated above the diaphragmatic hiatus to the carina level, in order to evaluate possible migration flows of the gastric remnant as reported in recent publications in this type of surgery.

All cases must be supervised by a radiologist as part of the study team to validate the images obtained with the purpose of being of the highest quality 3D for further processing. Validate the optimal degree of gastric distension. The data collected and stored in DICOM format for further manipulation 3D.

The study protocol provides for the realization of three CT scans:

1. Preoperative CT Be assessed the maximum gastric volume and the height of the esophagogastric junction in order to quantify the possible migration.
2. CT one month after surgery Possible to quantify the volume of gastric remnant and assess whether it has increased in volume. This data would adjust the actual volume of the remnant and apply it to the 3D model. Assess whether there is cranial migration of esophagogastric junction and gastric any late postoperative complications. Will correlate with weight loss.
3. CT one year after surgery Rating final state of the stomach, final quantification of the residual volume and correlation with final weight loss. Final assessment of the possible complications and gastric migration.

   * Scintigraphic evaluation Methodology

<!-- -->

1. Patient preparation It is important for the patient a 12 hours fast, to ensure that the stomach is empty. In addition, the patient may not smoke or take medication that could interfere with gastric motility. In diabetic patients, the CT scan wil be performed first thing in the morning, after the injection of insulin.
2. Radiopharmaceutical To get the most information in a single tracer, it is best to mark the solid component. With solids, in addition to assessing antral motility is measured indirectly by the state of the gastric tone, once they have been crushed and can be emptied. For this, 50 g huevina will beat with 1 mCi (37 MBq) of 99m Tc-sulfur colloid and immediately cook a tortilla.
3. Gamma camera Dual-head with low-energy collimator and medium resolution (LEAP)
4. Procedure Immediately after ingesting the food (in less than 10 minutes), it will proceed to detect of the stomach with the patient standing. Among the various detections, the patient should remain seated.

   Will immediately perform a baseline image and subsequently post-ingestion, anterior and posterior views of 2 minutes duration every 15 minutes for two hours.
5. Processed ROI is drawn over the gastric area, except in the first image to be included in all activity, even if there is intestinal.

   The software determines gastric accounts every time and projection (anterior and posterior) and geometric mean (Qty * Cpost). Also determined for each point the residual percentage compared to the initial activity.

   Time There will be temporary in the same sequence as in the radiological evaluation: preoperative and postoperative assessment at one month and a year
   * Functional esophagogastric evaluation Methodology Esophageal manometry and pH monitoring will be performed in all patients included in the study . The tests were carried out in the Digestive Pathology Service from Hospital Santa Creu i Sant Pau.

   Esophageal manometry catheter is made with a polyvinyl four holes spaced 5 inches between them. The distal end is connected to an external pressure transducer and the electrical signal is processed and analyzed by the computer program (PC Polygraf , Synectics Medical).

   It takes eight hours prior fasting , previously suspending medication that may alter esophageal motility and modifying stomach acid secretion.

   The catheter is inserted through the mouth into four channels that have reached the stomach. Recording the intra- gastric pressure at the end of expiration and is used as reference.

   The manometric evaluation of the lower esophageal sphincter is performed by a slow withdrawal. Record the resting pressure, length, location relative to the nasal ala and relaxation post swallow .

   Esophageal motor activity (amplitude and duration of the waves, peristaltic waves percentage of simultaneous post swallow), is evaluated by slowly withdrawn after conducting at least 10 swallows 3-5 cc of water every 20 seconds.

   Finally, we evaluate the upper esophageal sphincter activity. Pharyngeal pressure is recorded, the resting pressure of the upper esophageal sphincter pharyngo - esophageal coordination and upper esophageal sphincter relaxation after dry or liquid swallows every 20 seconds.

   After esophageal manometry pH monitoring is performed . Using a single-use probe 2 channels.

   We introduce the probe pH monitoring through the nose to reach the lower esophageal sphincter ( by reference to the location of the lower esophageal sphincter by manometry found). Probe is then removed, leaving 5 cm above the lower esophageal sphincter . The patient is instructed to perform their usual daily activity, a symptom diary recording . The probe is connected to a Holter apparatus that recorded during 24 the number of reflows , measure their duration in minutes and the duration of the longest reflux episode, the percentage of time that esophageal pH is less than 4. All measurements were recorded at both the proximal and distal esophagus. After 24 hours the tube is removed and information is processed by a computer program (PC Polygraf, Synectics Medical).

   Time The evaluation was conducted in three stages: pre-and postoperative assessment (within 2 days, 3 months and one year).

   - Hormonal and glucose metabolism

   It will carry out the following hormonal determinations:

   • Insulin

   • Glucagon

   • GLP-1

   • GIP

   • Ghrelin

   • Leptin

   • Adiponectin
   * Peptide YY

   Methodology Blood samples were made a week before surgery (in the Day Hospital of Endocrinology), during admission in ward General Surgery (on the 2nd postoperative day) and at 3 months and one year after surgery (in the Day Hospital of Endocrinology). To this end, each patient was placed in a peripheral vein upper extremity.
   * The first draw will be fasting.

   Ten minutes later, given a standard meal and proceed to the extraction of blood samples at the following times:
   * the end of the intake
   * postprandial samples (at 20, 60 and 120 respectively).

   Times:

   The determinations were carried out:
   * one week before surgery
   * postoperative day 2
   * a year

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years and less than 65 years
* BMI more than 40 kg/m2 or more than 35 kg/m2 with comorbidities likely to improve after weight loss.
* Morbid obesity established at least five years.
* Continued failures to adequately supervised conservative treatments
* Absence of endocrine disorders that are due to morbid obesity.
* Psychological stability:

  * No alcohol or drug abuse.
  * Absence of major psychiatric disorders (schizophrenia, psychosis), mental retardation, eating disorders (bulimia nervosa).
* Ability to understand the mechanisms to lose weight with surgery and understand that not always achieved good results.
* Understand that the goal of surgery is to achieve the ideal weight.
* Commitment for Adherence to surveillance guidelines after surgery
* Informed consent after receiving all the necessary information (oral and written).
* Women of childbearing age should avoid pregnancy for at least the first year after surgery

Exclusion Criteria:

* No acceptance
* Age less than 18 years or more than 65 years
* Previous bariatric surgery
* Previous gastric surgery
* Inflammatory bowel disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Body mass index | 1 year
Gastric volume | 1 month and 1 year

SECONDARY OUTCOMES:
Gastric emptying time | 1 year
Lower esophageal sphincter pressure | 1 year
Number of gastroesophageal reflux episodes | 1 year

OTHER OUTCOMES:
Hormone levels | 1 year
  Insulin, Glucagon, glucagon-like peptide (GLP-1), gastric inhibitory peptide (GIP), Ghrelin, Leptin, Adiponectin, Peptide YY

CONTACTS AND LOCATIONS:
Overall Officials: Maria Carmen Balagué Ponz, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Calle EE, Rodriguez C, Walker-Thurmond K, Thun MJ. Overweight, obesity, and mortality from cancer in a prospectively studied cohort of U.S. adults. N Engl J Med. 2003 Apr 24;348(17):1625-38. doi: 10.1056/NEJMoa021423. PMID 12711737
- [Background] Blackburn GL, Hutter MM, Harvey AM, Apovian CM, Boulton HR, Cummings S, Fallon JA, Greenberg I, Jiser ME, Jones DB, Jones SB, Kaplan LM, Kelly JJ, Kruger RS Jr, Lautz DB, Lenders CM, Lonigro R, Luce H, McNamara A, Mulligan AT, Paasche-Orlow MK, Perna FM, Pratt JS, Riley SM Jr, Robinson MK, Romanelli JR, Saltzman E, Schumann R, Shikora SA, Snow RL, Sogg S, Sullivan MA, Tarnoff M, Thompson CC, Wee CC, Ridley N, Auerbach J, Hu FB, Kirle L, Buckley RB, Annas CL. Expert panel on weight loss surgery: executive report update. Obesity (Silver Spring). 2009 May;17(5):842-62. doi: 10.1038/oby.2008.578. Epub 2009 Feb 19. PMID 19396063
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Regan JP, Inabnet WB, Gagner M, Pomp A. Early experience with two-stage laparoscopic Roux-en-Y gastric bypass as an alternative in the super-super obese patient. Obes Surg. 2003 Dec;13(6):861-4. doi: 10.1381/096089203322618669. PMID 14738671
- [Background] Alva S, Eisenberg D, Duffy A, Roberts K, Israel G, Bell R. Virtual three-dimensional computed tomography assessment of the gastric pouch following laparoscopic Roux-Y gastric bypass. Obes Surg. 2008 Apr;18(4):364-6. doi: 10.1007/s11695-008-9438-6. Epub 2008 Feb 15. PMID 18274830
- [Background] Karcz WK, Kuesters S, Marjanovic G, Suesslin D, Kotter E, Thomusch O, Hopt UT, Felmerer G, Langer M, Baumann T. 3D-MSCT gastric pouch volumetry in bariatric surgery-preliminary clinical results. Obes Surg. 2009 Apr;19(4):508-16. doi: 10.1007/s11695-008-9776-4. Epub 2008 Dec 18. PMID 19104904
- [Background] Melissas J, Koukouraki S, Askoxylakis J, Stathaki M, Daskalakis M, Perisinakis K, Karkavitsas N. Sleeve gastrectomy: a restrictive procedure? Obes Surg. 2007 Jan;17(1):57-62. doi: 10.1007/s11695-007-9006-5. PMID 17355769
- [Background] Braghetto I, Davanzo C, Korn O, Csendes A, Valladares H, Herrera E, Gonzalez P, Papapietro K. Scintigraphic evaluation of gastric emptying in obese patients submitted to sleeve gastrectomy compared to normal subjects. Obes Surg. 2009 Nov;19(11):1515-21. doi: 10.1007/s11695-009-9954-z. Epub 2009 Aug 28. PMID 19714384
- [Background] Shah S, Shah P, Todkar J, Gagner M, Sonar S, Solav S. Prospective controlled study of effect of laparoscopic sleeve gastrectomy on small bowel transit time and gastric emptying half-time in morbidly obese patients with type 2 diabetes mellitus. Surg Obes Relat Dis. 2010 Mar 4;6(2):152-7. doi: 10.1016/j.soard.2009.11.019. Epub 2009 Dec 22. PMID 20189465
- [Background] Bernstine H, Tzioni-Yehoshua R, Groshar D, Beglaibter N, Shikora S, Rosenthal RJ, Rubin M. Gastric emptying is not affected by sleeve gastrectomy--scintigraphic evaluation of gastric emptying after sleeve gastrectomy without removal of the gastric antrum. Obes Surg. 2009 Mar;19(3):293-8. doi: 10.1007/s11695-008-9791-5. Epub 2008 Dec 17. PMID 19089519
- [Background] Baumann T, Kuesters S, Grueneberger J, Marjanovic G, Zimmermann L, Schaefer AO, Hopt UT, Langer M, Karcz WK. Time-resolved MRI after ingestion of liquids reveals motility changes after laparoscopic sleeve gastrectomy--preliminary results. Obes Surg. 2011 Jan;21(1):95-101. doi: 10.1007/s11695-010-0317-6. PMID 21088924
- [Background] Pomerri F, Foletto M, Allegro G, Bernante P, Prevedello L, Muzzio PC. Laparoscopic sleeve gastrectomy--radiological assessment of fundus size and sleeve voiding. Obes Surg. 2011 Jul;21(7):858-63. doi: 10.1007/s11695-010-0255-3. PMID 20730606
- [Background] Parikh M, Eisner J, Hindman N, Balthazar E, Saunders JK. Tests of correlation between immediate postoperative gastroduodenal transit times and weight loss after laparoscopic sleeve gastrectomy. Surg Endosc. 2012 Dec;26(12):3548-51. doi: 10.1007/s00464-012-2352-y. Epub 2012 May 31. PMID 22648116
- [Background] Howard DD, Caban AM, Cendan JC, Ben-David K. Gastroesophageal reflux after sleeve gastrectomy in morbidly obese patients. Surg Obes Relat Dis. 2011 Nov-Dec;7(6):709-13. doi: 10.1016/j.soard.2011.08.003. Epub 2011 Aug 16. PMID 21955743
- [Background] Carter PR, LeBlanc KA, Hausmann MG, Kleinpeter KP, deBarros SN, Jones SM. Association between gastroesophageal reflux disease and laparoscopic sleeve gastrectomy. Surg Obes Relat Dis. 2011 Sep-Oct;7(5):569-72. doi: 10.1016/j.soard.2011.01.040. Epub 2011 Mar 22. PMID 21429818
- [Background] Braghetto I, Lanzarini E, Korn O, Valladares H, Molina JC, Henriquez A. Manometric changes of the lower esophageal sphincter after sleeve gastrectomy in obese patients. Obes Surg. 2010 Mar;20(3):357-62. doi: 10.1007/s11695-009-0040-3. Epub 2009 Dec 15. PMID 20013071
- [Background] Lazoura O, Zacharoulis D, Triantafyllidis G, Fanariotis M, Sioka E, Papamargaritis D, Tzovaras G. Symptoms of gastroesophageal reflux following laparoscopic sleeve gastrectomy are related to the final shape of the sleeve as depicted by radiology. Obes Surg. 2011 Mar;21(3):295-9. doi: 10.1007/s11695-010-0339-0. PMID 21165778
- [Background] Petersen WV, Schneider JH. Functional importance of laparoscopic sleeve gastrectomy for the lower esophageal sphincter in patients with morbid obesity. Obes Surg. 2012 Jun;22(6):949. doi: 10.1007/s11695-012-0612-5. No abstract available. PMID 22467053
- [Background] Chiu S, Birch DW, Shi X, Sharma AM, Karmali S. Effect of sleeve gastrectomy on gastroesophageal reflux disease: a systematic review. Surg Obes Relat Dis. 2011 Jul-Aug;7(4):510-5. doi: 10.1016/j.soard.2010.09.011. Epub 2010 Sep 21. PMID 21130052
- [Background] Gill RS, Birch DW, Shi X, Sharma AM, Karmali S. Sleeve gastrectomy and type 2 diabetes mellitus: a systematic review. Surg Obes Relat Dis. 2010 Nov-Dec;6(6):707-13. doi: 10.1016/j.soard.2010.07.011. Epub 2010 Aug 6. PMID 20947447
- [Background] Peterli R, Wolnerhanssen B, Peters T, Devaux N, Kern B, Christoffel-Courtin C, Drewe J, von Flue M, Beglinger C. Improvement in glucose metabolism after bariatric surgery: comparison of laparoscopic Roux-en-Y gastric bypass and laparoscopic sleeve gastrectomy: a prospective randomized trial. Ann Surg. 2009 Aug;250(2):234-41. doi: 10.1097/SLA.0b013e3181ae32e3. PMID 19638921